CLINICAL TRIAL: NCT02116920
Title: Evaluation of the Diagnostic Performance of HPV E6/E7 mRNA Versus Oncogenic HPV DNA as a Secondary Triage Test for VIA Positive Women in Cervical Cancer Screening Program
Brief Title: HPV E6/E7 mRNA Versus HPV DNA as Triage for Cervical Cancer Screening
Acronym: PODBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, Dr Sharmila Pimple, Professor in Preventive Oncology, Tata Memorial Hospital
Other Study IDs: BT/PR6121/SPD/11/1401/2012
Record Dates: First submitted 2014-03-25; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: CIN; Cervix Cancer
Keywords: CIN; HPV DNA; mRNA E6/E7; CIN triage; Cervix Biopsy; VIA; Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical Biopsy and Endo-cervical Brushing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VIA Positive: Those patients having acetowhite lesion over cervix on visual inspection after application of acetic acid

SUMMARY:
AIM: To develop and standardize a cost effective methodology or algorithm for mRNA E6/E7 for HPV genotypes 16, 18, 31, 33 and 45 as compared to commercially available assays which can be incorporated to triage excess false positives from primary screening for cervical cancers

Objectives:

1. Development and standardization of methodology /algorithm for mRNA E6/E7 testing for HPV genotypes 16, 18, 31, 33 and 45 using Real-time RT-PCR, in cervical samples.
2. To compare the test performance of this HPV E6/E7 mRNA assay to HPV DNA by HC 2 as secondary screening test, with the reference standard of colposcopy with biopsy, to triage women found positive in primary screening by VIA , in a population based screening for cancer of cervix.
3. To determine number of false positives in the primary screening test after testing VIA positives with a known high specificity secondary screening test (HPV-DNA HC II ) compared to HPV E6/E7 mRNA testing.

Study Population: Women in the age group of 30-65 years, who test positive on primary cervical screening test VIA will be enrolled for the proposed diagnostic tests along with reference standard of colposcopy with guided biopsy.

Methodology:

Women in the age group of 30-65 years undergoing routine cervical cancer screening through hospital ( Preventive Oncology screening clinic) and community based screening programs with abnormal test result using the primary cervical cancer screening test VIA will be recruited in the study. The primary screening test VIA will be administered by application of 5% Acetic Acid to the cervix and visualizing the cervix with the help of a halogen focus lamp. VIA will be considered to be positive if definite acetowhite lesions are visualized close to the squamocolumnar junction.

DETAILED DESCRIPTION:
AIM: To develop and standardize a cost effective methodology or algorithm for mRNA E6/E7 for HPV genotypes 16, 18, 31, 33 and 45 as compared to commercially available assays which can be incorporated to triage excess false positives from primary screening for cervical cancers.

Objectives:

1. Development and standardization of methodology /algorithm for mRNA E6/E7 testing for HPV genotypes 16, 18, 31, 33 and 45 using Real-time RT-PCR, in cervical samples.
2. To compare the test performance of this HPV E6/E7 mRNA assay to HPV DNA by HC 2 as secondary screening test, with the reference standard of colposcopy with biopsy, to triage women found positive in primary screening by VIA , in a population based screening for cancer of cervix.
3. To determine number of false positives in the primary screening test after testing VIA positives with a known high specificity secondary screening test (HPV-DNA HC II ) compared to HPV E6/E7 mRNA testing.

Study Population: Women in the age group of 30-65 years, who test positive on primary cervical screening test VIA will be enrolled for the proposed diagnostic tests along with reference standard of colposcopy with guided biopsy.

Study Site: Women tested positive on primary screening test VIA with referrals for further diagnostic testing at TMH will be enrolled under the study for proposed diagnostic tests along with reference test at tertiary care facility , Dept. of Preventive Oncology, Tata Memorial Hospital in Mumbai.

Sample Size To detect statistically significant difference in the test characteristics with 95% confidence limits, 80 % statistical power and alpha =0.05, we require to have around 180 cases of cervical intraepithelial neolplasia in the study.

With a demonstrated prevalence of around 2% for detecting high grade CIN lesions from our urban and rural community based cervical screening programmes, we need to enroll around 9,000 women from population based cervical cancer screening, to get 180 cases of cervical intraepithelial neolplasia

Methodology:

Women in the age group of 30-65 years undergoing routine cervical cancer screening through hospital ( Preventive Oncology screening clinic) and community based screening programs with abnormal test result using the primary cervical cancer screening test VIA will be recruited in the study. The primary screening test VIA will be administered by application of 5% Acetic Acid to the cervix and visualizing the cervix with the help of a halogen focus lamp. VIA will be considered to be positive if definite acetowhite lesions are visualized close to the squamocolumnar junction.

Criteria for a positive VIA test are presented below:

Positive VIA test:

1. Opaque, dense, dull, definite, well defined aceto white lesions, touching the squamocolumnar junction or close to the external os.
2. Strikingly dense acetowhite areas in the columnar epithelium.
3. Condyloma and Leukoplakia occurring closer to the squamocolumnar junction turning intensely white after application of acetic acid.
4. Growth on the cervix turning acetowhite.

The screened women who are tested Screen Positive by the primary screening test VIA will become eligible for recruitment in the study . Screen positive women from the outreach community screening programs will be referred to TMH ( Preventive Oncology screening clinic) for further diagnostic verification.

Participant Recruitment

The study participants will be recruited from Hospital ( Preventive Oncology screening clinic) and community based screening programmes in Mumbai. Medical Social Workers will explain the details and the purpose of the study to participants attending the screening clinic. Apparently healthy women in the age group of 30-65 yrs with an intact uterus and no past history of cervical neoplasia will become eligible to participate in the programme. If they are fulfilling the inclusion criteria given above, a written informed consent in the vernacular language (either Hindi or Marathi) will be obtained from the participant and a unique participant identification number will be assigned to the eligible women. Information on socio demographic and reproductive variables will then be collected using a detailed questionnaire.

Demographic, reproductive and sexual history data will be recorded at screening following informed consent..

Screen positive women will be tested for the presence of oncogenic HPV types by Hybrid Capture-II (HC-II) and HPV E6/E7 mRNA testing as diagnostic test. In addition to the above two tests all the screen positive women will also further receive Colposcopy with guided cervical biopsy, the reference gold standard test.

Colposcopy will be performed by trained doctors and the colposcopy impression will be noted down along with a punch biopsy from the aceto white area on the cervix detected by the primary screening test VIA. Biopsy specimens will be fixed in 10% formalin and will be processed and reported by the pathology laboratory at the Tata Memorial Centre.

The reference standard for final disease status will be histology.

Post Test Counseling :

At the end of all testing procedures post test counseling will be done by the Doctor and Medical Social Worker to explain the significance and the results of the testing procedures performed. The importance of follow up visit to understand the results of HPV/ mRNA E6/E7 and cervical biopsy will be explained to the women.

Follow up and Treatment:

Treatment for opportunistic and reproductive tract infections (RTI) will be provided. Women with High grade lesions (cervical precancers ) HSIL will be recommended to seek treatment with cryotherapy or LEEP (Loop Electrosurgical Excision Procedure) or by cold knife conization at the Tata Memorial Centre Mumbai.

Total Project Period: Three years:

Proposal submission, training, participant recruitment, data collection and analysis, including follow-up of cases at the end of enrollment period

ELIGIBILITY:
Inclusion Criteria:

1. Female between 30-65years of age
2. Not pregnant by menstrual history
3. No history of prior treatment for cancer of the cervix
4. No history of hysterectomy
5. Healthy enough to undergo a pelvic examination, i.e., not seriously ill with a debilitating condition

Exclusion Criteria:

1. Women below and above this age group
2. Women already screened and detected for cervical precencers and cancers
3. Women with debilitating condition
4. Women with Hysterectomy
5. Women whom are pregnant

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in the age group of 30 to 65 years (non pregnant and with intact uterus) in urban slum colonies of Mumbai city
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome Measure | 3 Years
  Sensitivity and specificity of HPV DNA test versus E6/E7 mRNA test against gold standard of histopathology confirmed CINs.
  After the above mentioned time frame, efficacy of 1. HPV DNA Test and 2. E6/E7 mRNA test will be evaluated.
  Such evaluation is not applicable for individual participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila A Pimple, Professor, Principal Investigator — TMH, Tata Memorial Centre, Mumbai; Tanuja R Teni, SciOfficerF, Principal Investigator — ACTREC, Tata Memorial Centre, Mumbai; Gauravi A Mishra, Assoc Prof, Principal Investigator — TMH, Tata Memorial Centra, Mumbai; Surendra S Shastri, HOD, Principal Investigator — TMH, Tata Memorial Centre, Mumbai
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- See also: Tata Memorial Centre, Mumbai web site — http://tmc.gov.in